CLINICAL TRIAL: NCT01438398
Title: A Prospective, Single Center, Proof of Concept Pilot Study of the Efficacy and Safety of Submucosal Endoscopic Myotomy With Mucosal Flap (SEMF) Technique in the Treatment of Patients With Achalasia
Brief Title: Efficacy & Safety of Submucosal Endoscopic Myotomy With Mucosal Flap (SEMF) in the Treatment of Patients With Achalasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, Stavros Stavropoulos, MD, Advanced Endoscopist, Winthrop University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10035
Record Dates: First submitted 2011-03-28; First posted 2011-09-22 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Achalasia; Dysphagia
Keywords: Submucosal endoscopic myotomy; Per Oral Endoscopic Myotomy; Natural Orifice Transluminal Endoscopic Surgery
MeSH Terms: conditions — Esophageal Achalasia; Deglutition Disorders | interventions — Natural Orifice Endoscopic Surgery; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Submucosal Endoscopic Mucosal Flap Technique (Other): Submucosal Endoscopic Mucosal Flap Technique
  Interventions: Procedure: Submucosal endoscopic myotomy with mucosal flap technique; Procedure: Submucosal Endoscopic Mucosal Flap (SEMF) technique

INTERVENTIONS:
Procedure: Submucosal endoscopic myotomy with mucosal flap technique — Submucosal Endoscopy with Mucosal Flap (SEMF) technique involves the following: (1) injecting 0.9 % normal saline solution to create a submucosal cushion, (2) tiny cut is made into the cushion, (3) Balloon will be used to dilate the opening and allow passage of endoscope in the submucosal space, (4) Upon direct visualization of the muscle fibers, the doctor will cut the circular layers of the diseased muscles, and (5) Tiny clips will be used to close the tiny cut made earlier.
  Other Names: Per Oral Endoscopic Myotomy (POEM); Natural Orifice Transluminal Endoscopic Surgery (NOTES)
Procedure: Submucosal Endoscopic Mucosal Flap (SEMF) technique
  Other Names: Per Oral Endoscopic Myotomy; Natural Orifice Transluminal Endoscopic Surgery

SUMMARY:
The purpose of this study is to learn about the safety and usefulness of a procedure called endoscopic submucosal myotomy, which is a new technique in the treatment of achalasia. Achalasia is a disorder involving the lack of smooth muscle relaxation and sustained high pressure in the sphincter (muscle) of the lower esophagus. This may result in symptoms such as difficulty in swallowing, chest pain, regurgitation of food and eventually, weight loss.

For more than a decade, a laparoscopic surgical procedure known as Heller myotomy has been the primary treatment for achalasia in patients with low surgical risk. In Heller myotomy, the surgeon makes three to four small abdominal incisions, inserts tube-like instruments through them, and once inside, the junction between the esophagus and stomach is found, a lengthwise incision is made on the muscular ring surrounding the lower esophageal sphincter which weakens the muscle and the lower esophageal sphincter or muscle (LES) is then able to open more easily. However, there is an emerging field known as natural orifice (opening) transluminal (through the lumen) endoscopic surgery (NOTES). This approach involves passing an endoscope - a thin tube with a built-in camera, light and minuscule tools through the natural opening in the body, like the mouth in order to perform less invasive surgery without any external wounds or scars. The procedure is done using the Submucosal Endoscopy with Mucosal Flap (SEMF) technique which involves passing an endoscope through the mouth into the esophagus, where a small incision is made on the lining of the esophagus, known as the mucosa. A balloon is then inserted and dilated in the submucosa - the layer between the inner lining of the esophagus and the outer wall consisting of the muscle of the esophagus. Dilation of the balloon in the submucosa creates a tunnel that allows insertion of the endoscope and access to the muscle of the lower esophageal sphincter (LES). A long incision is then carefully made on the posterior portion of the muscular ring that forms the LES. The incision divides the muscle fibers of the LES, which weakens the muscle, allowing for the easier passage of food while preserving some valve function to prevent reflux of acid from the stomach into the esophagus.

The expected duration of participation is up to 10 years from the time study participants undergo the endoscopic surgical procedure.

DETAILED DESCRIPTION:
The safety of the procedure and feasibility of the study will be measured by improvement in subjects' symptoms score, decrease in LES pressure, as well as the number and severity of complications or adverse events experienced by the subjects. A modified Eckhardt dysphagia assessment tool will be used in grading the dysphagia symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older, male or female, belonging to any race or ethnic origin
2. Patients with manometric positive diagnosis of achalasia, with corresponding symptoms of dysphagia, regurgitation of food or chest pain
3. Patients who are willing and competent to sign Informed Consent and to comply with study related visits and procedures

Exclusion Criteria:

1. Patients who are below 18 years of age
2. Presence of coagulopathy
3. Pregnancy
4. Patients who, in the investigator's opinion, are medically unstable, are unable to give informed consent, or whose risks outweigh the benefits of participating in the study
5. Vulnerable subjects: Prisoners, persons with decisional incapacity, and any person who are directly involved in the study, including their immediate family members, and anybody who may have any conflict of interest such as employees of ERBE, USA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-04-08 (Actual); Primary Completion 2015-01-06 (Actual); Study Completion 2015-10-22 (Actual)

PRIMARY OUTCOMES:
Change in Lower esophageal sphincter pressure (LES) | at 3 months post endoscopic myotomy
  High Resolution Esophageal Manometry will be done at 3 months to measure LES and the result will be compared to baseline or pre-endoscopic myotomy LES pressure.
Change in frequency of dysphagia | 4 weeks post procedure
  Swallowing difficulty (dysphagia) will be assessed using the Modified Eckhardt Dysphagia Assessment Tool which includes asking the patient how often he/she experiences swallowing difficulty (0 = none, 1 = occasional, 2 = daily, and 3 = every meal. The score will be compared to pre-myotomy score.
Change in frequency of Regurgitation | 4 weeks post procedure
  Patient will be asked how often he/she brings up swallowed liquid/solid food or regurgitates (0 = none, 1 = occasional, 2 = daily, and 3 = every meal. The score will be compared to the score prior to the procedure.
Change in frequency of chest pain | 4 weeks post procedure
  The patient will be asked how often he/she experiences chest pain and the frequency (0 = none, 1 = occasional, 2 = daily, and 3 = every meal. The score will be compared to pre-myotomy score.
Presence of perforation | During endoscopic myotomy procedure
  Presence of perforation that is seen during the endoscopic procedure.
Presence of bleeding | During endoscopic myotomy procedure
  Occurence of bleeding during the procedure.
Presence of mediastinal emphysema | During endoscopic myotomy procedure
  Presence of mediastinal emphysema will be recorded.
Presence of Infection | 4 weeks post procedure
  Presence of infection within the first 4 weeks post myotomy will be recorded.
Development of stricture at the myotomy site. | 3 months post procedure
  Development of stricture will be assessed by performing an upper endoscopy for patients with change in their Modified Dysphagia Score.

SECONDARY OUTCOMES:
Presence and frequency of heartburn | 4 weeks post procedure
  The patient will be asked for presence or absence of heartburn. If present, he/she will be asked for frequency (0 = none, 1 = occasional, 2 = daily, and 3 = every meal). The score will be compared to pre-myotomy score.
Frequency of use of antacids (PPI, H-2 antagonists) | 4 weeks post procedure
  The patient will be asked if he/she is using any type of antacid. If using antacid, he/she will be asked how often he/she is using it (0 = none, 1 = occasional, 2 = daily, and 3 = every meal). The score will be compared to pre-myotomy score.
Change in patient's weight | At 3, 6, 9, and 12 months post procedure.
  Post myotomy weight will be measured and recorded and compared to pre-myotomy weight.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros N Stavropoulos, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States